CLINICAL TRIAL: NCT02135263
Title: Metabolism of Methylphenidate and Enalapril Based on CES1 Genotype
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Mental Health Centre Sct. Hans (Denmark) (Unknown); University of Copenhagen (Other); The Leiden Academic Center for Drug Research (LACDR) (Unknown); Duke University (Other)
Responsible Party: Principal Investigator, Gesche Jurgens, M.D., Ph.D., Bispebjerg Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INDICES-WP2
Record Dates: First submitted 2013-07-01; First posted 2014-05-09 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Carboxylesterase 1 (CES1) Genotype; CES1 Activity
MeSH Terms: interventions — Methylphenidate; Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate
- Enalapril (Experimental)
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Methylphenidate — 10 mg as a single dose followed by blood samples for the next 33 hours
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Enalapril — 10 mg as a single dose followed by blood samples for the next 72 hours
  Other Names: Corodil
  Arms: Enalapril

SUMMARY:
The purpose of this study is to determine whether differences in the gene coding for the liver enzyme carboxylesterase 1 (CES1) means differences in the metabolism of two CES1 dependent drugs, enalapril and methylphenidate.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Caucasian

Exclusion Criteria:

* Chronic disease (except hay fever and eczema)
* Pregnancy
* Smoking
* High level of alcohol consumption (> 21 units per week for men and 14 for women)
* Known allergy towards methylphenidate and enalapril
* Permanent use of medication (contraception ok)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of methylphenidate | Predose, ½, 1, 1½, 2, 2½, 3, 4, 6, 8, 10, 24 and 33 hours post-dose
Time to peak plasma concentration (Tmax) of methylphenidate | Predose, ½, 1, 1½, 2, 2½, 3, 4, 6, 8, 10, 24 and 33 hours post-dose
Terminal half life (t½) of methylphenidate | Predose, ½, 1, 1½, 2, 2½, 3, 4, 6, 8, 10, 24 and 33 hours post-dose
Area under the plasma concentration versus time curve (AUC) of methylphenidate | Predose, ½, 1, 1½, 2, 2½, 3, 4, 6, 8, 10, 24 and 33 hours post-dose
Peak plasma concentration (Cmax) of enalapril | Predose, ½, 1, 2, 3, 4, 5, 6, 9, 24, 48 and 72 hours post-dose
Time to peak plasma concentration (Tmax) of enalapril | Predose, ½, 1, 2, 3, 4, 5, 6, 9, 24, 48 and 72 hours post-dose
Terminal half life (t½) of enalapril | Predose, ½, 1, 2, 3, 4, 5, 6, 9, 24, 48 and 72 hours post-dose
Area under the plasma concentration versus time curve (AUC) of enalapril | Predose, ½, 1, 2, 3, 4, 5, 6, 9, 24, 48 and 72 hours post-dose

SECONDARY OUTCOMES:
Metabolomic profile | Predose/pre-meal, predose/post-meal, 2 and 6 hours post-dose
  Four samples for each participant during the methylphenidate trials (as indicated above). Metabolomics will be assessed with focus on lipids (lipid platform) and with use of usual concentration measures (eg nanomolar (nM))

CONTACTS AND LOCATIONS:
Overall Officials: Gesche Jürgens, M.D., Principal Investigator — Department of Clinical Pharmacology, Bispebjerg University Hospital
Locations (1):
- Department of Clinical Pharmacology, Bispebjerg University Hospital, Copenhagen, Denmark